CLINICAL TRIAL: NCT05005091
Title: Effect of Preoperative Oral Carbohydrate Administration in Thoracic Surgery
Brief Title: Effect of Preoperative Oral Carbohydrate Administration in Thoracic Surgery Patients
Acronym: oralcarbohydra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cansel Atinkaya Baytemir, SureyyapasaM, Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SureyyapasaM
Record Dates: First submitted 2021-08-08; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Non Small Cell Lung Cancer; Fasting; Postoperative Pneumonia
Keywords: Preoperative fasting, postoperative morbidity, preoperative carbohydrate drinking, thoracic surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Fasting | interventions — Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral carbohydrate (Active Comparator): the patients drunk oral carbohydrate two hours ago preoperatively
  Interventions: Dietary Supplement: Oral carbohydrate
- no oral carbohydrate (No Intervention): the patients did not drink oral carbohydrate preoperatively

INTERVENTIONS:
Dietary Supplement: Oral carbohydrate — 100 ml oral carbohydrate two hours ago preoperatively
  Arms: oral carbohydrate

SUMMARY:
Preoperative carbohydrate loading has been shown to reduce pre-operative discomfort and postoperative nausea and vomiting. There is no need for prolonged preoperative fasting of the patients, but the traditional approach still continues especially in thoracic surgery patients. For this purpose, we aimed to evaluate the effect of preoperative carbohydrate loading on postoperative morbidity in the patients.

DETAILED DESCRIPTION:
The study was conducted on 94 patients. The patients in the control group were fasting after midnight. Experimental group patients consumed carbohydrate drink as liquid two hours before the operation. 47 patients were in the control group (A) and 47 patients were in the experimental group (B). The groups were compared in terms of length of hospital and intensive care unit stay, vomiting, gas-stool outlet, postoperative pain conditions (VAS), inflammation parameters, blood glucose, and mobilization time.

SPSS 11.0 (SPSS, Inc., Chicago, IL, USA) was used for statistical analyses. All means were presented with 95% confidence limits. In the empirical analysis, t-test and chi-square test were used. In addition, correlation analysis was used to determine the relationship between fasting time and surgical recovery time.

ELIGIBILITY:
Inclusion Criteria:

Stage I-Stage II all operable NSCLC patients -

Exclusion Criteria:

Patients with diabetes mellitus, a history of delayed gastric emptying, severe hepatic or renal failure, or any endocrine disorder that might influence the metabolic parameters were excluded, as were patients requiring urgent or emergent surgery.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Mobilization time | 1 hour
  postoperative mobilization

CONTACTS AND LOCATIONS:
Locations (1):
- health Science University, Sureyyapa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No